CLINICAL TRIAL: NCT02156076
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Arm Study to Evaluate the Safety, Tolerability, and Effect on Atrial Fibrillation Burden of BMS-919373 in Patients With Paroxysmal Atrial Fibrillation
Brief Title: A Blinded Study to Evaluate Effect on Atrial Fibrillation Burden in Patients With Paroxysmal Atrial Fibrillation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on business reasons, unrelated to safety
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CV205-005
Record Dates: First submitted 2014-05-12; First posted 2014-06-05 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: Placebo (Matching with BMS-919373) (Placebo Comparator): Placebo (Matching with BMS-919373) 0 mg tablets orally once daily for approximately 28 Days
  Interventions: Drug: Placebo (Matching with BMS-919373)
- Arm B: BMS-919373 (Experimental): BMS-919373 3 mg tablets orally once daily for approximately 28 days
  Interventions: Drug: BMS-919373
- Arm C: BMS-919373 (Experimental): BMS-919373 5 mg tablets orally once daily for approximately 28 days
  Interventions: Drug: BMS-919373
- Arm D: BMS-919373 (Experimental): BMS-919373 12 mg tablets orally once daily for approximately 28 days
  Interventions: Drug: BMS-919373

INTERVENTIONS:
Drug: BMS-919373
  Arms: Arm B: BMS-919373; Arm C: BMS-919373; Arm D: BMS-919373
Drug: Placebo (Matching with BMS-919373)
  Arms: Arm A: Placebo (Matching with BMS-919373)

SUMMARY:
The purpose of this study is to evaluate the effect of BMS-919373 on atrial fibrillation (AF) through its effect on AF burden (AFB), or the percent of time in AF, in subjects with paroxysmal AF (pAF) when administered orally at a range of doses (2 mg once daily (QD), 5 mg QD, 12 mg QD following a 1-week period of loading doses of 3 mg QD, 8 mg QD and 20 mg QD, respectively) for a total of 4 weeks. It is hypothesized that treatment with BMS-919373 will reduce AF burden as compared to baseline relative to placebo.

DETAILED DESCRIPTION:
Primary Purpose: Protocol designed to assess, by the use of long term non-invasive beat-to-beat monitoring with the SEEQ Mobile Cardiac Telemetry (MCT) system, the effect of BMS-919373 on the percent change from baseline relative to placebo of atrial fibrillation burden in subjects with paroxysmal atrial fibrillation.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Signed informed consent
* Paroxysmal Atrial Fibrillation (pAF) with available documentation of AF and reporting symptoms within 6 months prior to screening
* Able to tolerate withdrawal of antiarrhythmic therapy (rhythm control)
* Echocardiographically measured left ventricular ejection fraction (LVEF) ≥40%,measured within 12 months of enrollment
* Echocardiographically measured left atrial (LA) diameter ≤ 5.0 cm, measured within 12 months of enrollment

Exclusion Criteria:

* Women of childbearing potential
* AFB < 3% or > 70%, during both screening periods independently
* Permanent or persistent Atrial Fibrillation
* Cardioversion within 3 months of study drug administration
* Stroke within 12 months of study drug administration
* TIA within 12 months of study drug administration
* Heart failure of NYHA class III or greater (symptoms of heart failure at rest or with minimal exertion)
* Heart failure of NYHA class II (symptoms of heart failure with routine levels of exertion)with ejection fraction <40% as measured by echocardiography at any time within 12 months of study enrollment (i.e. additional ejection fraction measurements ≥ 40% over this period will not counter this exclusion)
* Valvular heart disease (including any valvular insufficiency or stenosis greater than"mild")
* Ablation within 3 months of study enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (19):
  - Cardiology Consultants Of Orange County Med. Group Inc, Anaheim, California
  - Oracle Clinical Research, Inc., Anaheim, California
  - Wcct Global, Llc, Costa Mesa, California
  - Long Beach Va Medical Center, Long Beach, California
  - Spectrum Clinical Research, Moreno Valley, California
  - Chase Medical Research, Llc, Waterbury, Connecticut
  - All Medical Research, Llc, Cooper City, Florida
  - The Cardiac And Vascular Institute Research Foundation, Llc, Gainesville, Florida
  - Acrc Cardiology, Lake Worth, Florida
  - The Heart Institute At Largo, Largo, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Community Clinical Research Center, Anderson, Indiana
  - Midwest Heart And Vascular Specialists, Llc., Overland Park, Kansas
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Castlerock Clinical Research Consultants, Llc, Tulsa, Oklahoma
  - Capital Area Research, Llc, Camp Hill, Pennsylvania
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - Local Institution, Austin, Texas
  - Utah Cardiology P.C, Layton, Utah
- Canada (14):
  - Local Institution, Edmonton, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - Local Institution, Cambridge, Ontario
  - Dr. Andy S.C. Lam Medicine Professional, Grimsby, Ontario
  - Stroke Prevention & Artherosclerosis Research Centre, London, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Oshawa, Ontario
  - King Street Cardiology, Oshawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Csss Du Sud De Lanaudiere-Hopital Pierre-Le Gardeur, Terrebonne, Quebec

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 158 participants were enrolled out of which 26 participants were randomized and treated.
Groups:
- BMS-919373 3/2 mg: Participants received loading dose of BMS-919373 3 milligram (mg) as oral tablets (each tablet of 1 mg*3) once daily (QD) for one week followed by maintenance dose of BMS-919373 2 mg as oral tablets (each tablet of 1 mg*2) QD for 3 weeks.
- BMS-919373 8/5 mg: Participants received loading dose of BMS-919373 8 mg as oral tablets (each tablet of 1 mg*3 + 5 mg*1) QD for one week followed by maintenance dose of BMS-919373 5 mg as oral tablets (each tablet of 5 mg*1) QD for 3 weeks.
- BMS-919373 20/12 mg: Participants received loading dose of BMS-919373 20 mg as oral tablets (each tablet of 5 mg*4) QD for one week followed by maintenance dose of BMS-919373 12 mg as oral tablets (each tablet of 5 mg*2 + 1 mg*2) QD for 3 weeks.
- Placebo: Participants received placebo matching with BMS-919373 0 mg tablets (4 tablets) orally QD for 28 Days.
Period: Treatment Period
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Started | 7 | 7 | 6 | 6
Completed | 7 | 5 | 4 | 4
Not Completed | 0 | 2 | 2 | 2
Not completed — no longer meets study criteria | 0 | 0 | 1 | 0
Not completed — Poor/non-compliance | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Subject request to discontinue treatment | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Follow-up Period
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Started | 7 | 5 | 4 | 4
Completed | 6 | 5 | 4 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 6 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (5.83) | 61.0 (8.23) | 65.7 (10.05) | 65.0 (10.77) | 65.4 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 2 | 7
  Male | 6 | 4 | 5 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 5 | 5 | 3 | 3 | 16
  Unknown or Not Reported | 2 | 1 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 7 | 7 | 4 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Atrial Fibrillation Burden (AFB) as Assessed by SEEQ Mobile Cardiac Telemetry (MCT) System
Description: AFB is defined as the percent of time spent in atrial fibrillation (AF). AFB will be assessed by use of long term non- invasive beat-to-beat monitoring with the SEEQ MCT system. This technology consists of a low-profile adhesive patch that has been approved for continuous use for up to 30 days. The patch is able to continuously record electrocardiographic signals and, in conjunction with a wirelessly connected portable cellular communications device, transmit these signals for real-time analysis, including atrial and ventricular arrhythmias and AFB.
Time Frame: Day 8 to Day 29
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-related AEs and Death
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product. A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect.
Time Frame: Up to Day 50
Population: All treated participants included all the participants who have received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants
  AEs | 4 | 4 | 3 | 4
  SAEs | 0 | 0 | 0 | 0
  Treatment-related AEs | 0 | 3 | 0 | 0
  Death | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Concentarion (Cmax) of BMS-919373
Description: Cmax is defined as the maximum observed concentration of BMS-919373.
Time Frame: Day 1 and Day 22: Predose 1, 2, and 4 hours postdose
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Trough Observed Concentration (Cmin) of BMS-919373
Description: Ctrough is defined as the minimum estimated plasma concentration at steady state.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Oral Clearance (CL/F) of BMS-919373
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Central Volume of Distribution (Vc/F) of BMS-919373
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug is uniformly distributed to produce the desired plasma concentration of a drug. Vc/F is a hypothetical volume into which a drug initially distributes upon administration.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Absorption Rate Constant (Ka) of BMS-919373
Description: Ka is the absorption rate constant.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Average Concentration (Cavg) of BMS-919373 at Steady State
Description: Cavg is defines as the average concentration at steady state.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Area Under the Concentration-time Curve (AUC) at Steady State of BMS-919373
Description: AUC is defined as the area under the concentration-time curve at steady state.
Time Frame: Day 8 (predose), Day 22 (predose, 1, 2, and 4 hours postdose), and Day 29 (24 hours after last dose of Day 28)
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Time to First Atrial Fibrillation Recurrence (TTFR) (Symptomatic or Asymptomatic)
Description: The TTFR is defined as the time to the first MCT-recorded AF episode after the first loading dose on Day 1. MCT will provide both "System-triggered" and "Patient-triggered" results and report them separately. "System-triggered" results will include both symptomatic and asymptomatic findings, while "Patient-triggered" results will be the symptomatic ones triggered to report by patients. The analysis will be done both for "System-triggered" and for "Patient-triggered" results.
Time Frame: Day 8 to Day 29
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Total Number of Atrial Fibrillation Episodes
Description: The total number AF episodes were derived from AF episode histogram data over the monitoring period.
Time Frame: Day 8 to Day 29
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Average Duration of Atrial Fibrillation Per Episode
Description: The average duration of AF per episode was calculated from the total time a participant in AF and the total number of AF episodes over the monitoring period.
Time Frame: Day 8 to Day 29
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 50 days
Description: All treated participants included all the participants who have received at least one dose of study treatment.
Arm/Group | Placebo | BMS-919373 3/2 mg | BMS-919373 8/5 mg | BMS-919373 20/12 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/7 | 4/7 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | BMS-919373 3/2 mg (N=7) | BMS-919373 8/5 mg (N=7) | BMS-919373 20/12 mg (N=6)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Energy Increased (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Medical Device Site Dermatitis (General disorders) | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0
Head Discomfort (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Choking Sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor decided to terminate development of BMS-919373 for business reasons unrelated to safety, due to which data was not analyzed for maximum outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.